CLINICAL TRIAL: NCT06050395
Title: The MONITOR Study: Remote Monitoring Of a Nutrition Intervention To Optimize Treatment Response
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-22523
Record Dates: First submitted 2023-09-11; First posted 2023-09-22 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MONITOR group: Monitoring of a Nutrition Intervention to Optimize treatment Response (Experimental): Participants randomized to the MONITOR arm will be provided dietary coaching biweekly to discuss nutrition concerns, anti-inflammatory diet compliance, and set SMART goals based on their most recent Vioscreen food frequency questionnaires.
  Interventions: Behavioral: Quality fo Life Questionnaire (FHSI); Behavioral: Vioscreen Food Frequency Questionnaire (FFQ); Behavioral: NutritionCoaching; Behavioral: Follow-Up Survey; Behavioral: Functional Assessment of Anorexia/Cachexia Treatment (FAACT) Questionnaire; Behavioral: Patient Reported Outcomes Measure- Cognitive Function (PROMIS-Cog) Questionnaire
- Standard Usual Care (Active Comparator): Standard Usual Care participants will receive usual nutrition care received in the Moffitt Cancer Center pancreatic clinic, in addition to handouts on diet.
  Interventions: Behavioral: Quality fo Life Questionnaire (FHSI); Behavioral: Educational Handouts; Behavioral: Follow-Up Survey; Behavioral: Functional Assessment of Anorexia/Cachexia Treatment (FAACT) Questionnaire; Behavioral: Patient Reported Outcomes Measure- Cognitive Function (PROMIS-Cog) Questionnaire

INTERVENTIONS:
Behavioral: Quality fo Life Questionnaire (FHSI) — Participants will take a survey at baseline and visit 2 (weeks 6-8), and visit 3 (week 10-14). The Functional Assessment of Cancer Therapy Hepatobiliary Cancer Symptom Index-8 (FHSI) questionnaire uses a 5-point Likert-type scale, 0=not at all and 4=Very much. A lower total score indicates better quality of life.
Behavioral: Vioscreen Food Frequency Questionnaire (FFQ) — Participants will receive a web-based link and information to complete VioScreen, a web-based food frequency questionnaire, which allows participants to choose the average frequency of consumption of food items over a given time frame (1 month, 3 month, 1 year, etc.) on a Likert scale with choices ranging by individual questions. Total energy and nutrient intake is estimated by summing intakes from each food based on the selected portion size, reported frequency of consumption, and nutrient content of each food item. Anti-inflammatory and pro-inflammatory dietary patterns are calculated using the energy-adjusted dietary inflammatory index (DII) score to represent the inflammatory potential of an individual's overall diet, using data from FFQ responses. Higher DII scores represent more pro-inflammatory diets while lower (i.e., more negative) DII scores represent more anti-inflammatory diet.
  Arms: MONITOR group: Monitoring of a Nutrition Intervention to Optimize treatment Response
Behavioral: Educational Handouts — Participants will receive educational handouts on diet.
  Arms: Standard Usual Care
Behavioral: NutritionCoaching — Participants will receive bi-weekly nutrition coaching on anti-inflammatory dietary patterns and foods.
  Arms: MONITOR group: Monitoring of a Nutrition Intervention to Optimize treatment Response
Behavioral: Follow-Up Survey — Participants will complete a custom exit/follow up survey regarding relevance, acceptability, intervention length and timing, an barriers/facilitators. This survey contains 38 questions scored from 1 -Strongly agree to 5-Strongly disagree. A lower score indicates patient satisfaction with the program and the skills and knowledge gained in the program.
Behavioral: Functional Assessment of Anorexia/Cachexia Treatment (FAACT) Questionnaire — The FAACT questionnaire uses a 5 point Likert-type scale, 0=Not at all, 4=Very much. A higher score indicates better appetite and quality of life.
Behavioral: Patient Reported Outcomes Measure- Cognitive Function (PROMIS-Cog) Questionnaire — Participants will complete the PROMIS-Cog form which measures self-reported cognitive deficits. The questionnaire uses a 5 point Likert-type scale, 1=Very often and 5=Never. A higher score indicates higher cognitive function.

SUMMARY:
The purpose of the study is to evaluate the feasibility and acceptability of a remote nutrition coaching and monitoring intervention during the 12-weeks of active chemotherapy for borderline resectable and locally advanced pancreatic cancer participants.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years of age or more
* Newly diagnosed, in place tumors of the pancreas
* No documented or observable psychiatric or neurological disorders that would interfere with study participation (e.g., dementia, psychosis)
* Able to speak and read English
* Able to consume food orally
* Chemotherapy naive
* Scheduled to receive treatment with chemotherapy
* Able to provide verbal informed consent

Exclusion Criteria:

* Women who are pregnant
* Pancreatic cancer not the primary diagnosis
* Patients on enteral or parental nutrition
* Patients with metastatic pancreatic cancer
* Patients with evidence of impeding bowel obstruction
* Patients presenting with ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2026-02-13 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate -Feasibility | Up to 8 months
  The study will be deemed feasible if >/= 60% of eligible participants are enrolled
Retention Rate - Feasibility | at 12 weeks
  The study will be deemed feasible if >/=70% of participants complete the post-intervention questionnaire
Adherence - Feasibility | at 12 weeks
  The study will be deemed feasible if average attendance is >/=4 weeks of sessions (out of 6) for MONITOR arm

SECONDARY OUTCOMES:
Participant Satisfaction with Overall Program- Acceptability | at 12 weeks
  The study will be deemed acceptable based on the satisfaction score on follow-up survey. The follow-up survey uses open-ended and likert-style questions regarding 1) relevance and applicability of the MONITOR intervention content and objective/subjective data collection methods; 2) intervention length and timing; and 3) barriers/facilitators to participation and retention. On a 5-point Lkert-type scale, a(1) =strongly agree and e(5)=strongly disagree. Participant Satisfaction with Overall Program is determined by a score >/=3 on a 5-point scale.
Participant intent to continue using skills- Acceptability | at 12 weeks
  The study will be deemed acceptable based on the satisfaction score on follow-up survey. The follow-up survey uses open-ended and likert-style questions regarding 1) relevance and applicability of the MONITOR intervention content and objective/subjective data collection methods; 2) intervention length and timing; and 3) barriers/facilitators to participation and retention. On a 5-point Lkert-type scale, a(1) =strongly agree and e(5)=strongly disagree. Participant intent to continue using skills- is determined by a score >/=3 on a 5-point scale.
Participant perception of utility of knowledge gained - Acceptability | at 12 weeks
  The study will be deemed acceptable based on the satisfaction score on follow-up survey. The follow-up survey uses open-ended and likert-style questions regarding 1) relevance and applicability of the MONITOR intervention content and objective/subjective data collection methods; 2) intervention length and timing; and 3) barriers/facilitators to participation and retention. On a 5-point Lkert-type scale, a(1) =strongly agree and e(5)=strongly disagree. Participant perception of utility of knowledge gained is determined by a score >/=3 on a 5-point scale.

OTHER OUTCOMES:
Treatment Effect - Quality of Life | at Baseline, and at 6 and 12 weeks
  Quality of Life will be measured using the FACT-Hep questionnaire. Participants will take the Functional Assessment of Cancer Therapy Hepatobiliary Cancer Symptom 8 Item Version (FHSI) questionnaire which uses a 5-point likert-type scale, 0=not at all and 4=Very much. A lower total score indicates better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Crowder, PhD, Principal Investigator — Moffitt Cancer Center; Pamela Hodul, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided